CLINICAL TRIAL: NCT07254390
Title: Effects of Trans-Auricular Vagal Stimulation on Neuromotor Recovery Post-Stroke in the Subacute Phase During Training With the Khymeia Technological Device and Traditional Rehabilitation
Brief Title: Effects of Trans-Auricular Vagal Stimulation on Neuromotor Recovery in Subacute Stroke During Technological and Traditional Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2665
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Transcutaneous vagus nerve stimulation (tVNS); Stroke rehabilitation; Neuroplasticity; Upper limb motor recovery; Non-invasive neuromodulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Khymeia + Active tVNS (Experimental)
  Interventions: Device: Active trans-auricular vagus nerve stimulation (tVNS) + Khymeia training
- Khymeia + Sham tVNS (Sham Comparator)
  Interventions: Device: Sham trans-auricular vagus nerve stimulation + Khymeia training
- Traditional Rehabilitation + Active tVNS (Experimental)
  Interventions: Device: Traditional Rehabilitation + Active tVNS
- Traditional Rehabilitation + Sham tVNS (Sham Comparator)
  Interventions: Device: Traditional Rehabilitation + Sham tVNS

INTERVENTIONS:
Device: Active trans-auricular vagus nerve stimulation (tVNS) + Khymeia training — Active trans-auricular vagus nerve stimulation (tVNS) with the Parasym® device (CE 0197). Electrode placed on the left tragus, 25 Hz, 250 µs, intensity to tolerance, 60 min/day, 5 days/week for 4 weeks, combined with Khymeia robotic upper limb rehabilitation.
  Arms: Khymeia + Active tVNS
Device: Sham trans-auricular vagus nerve stimulation + Khymeia training — Sham tVNS using the Parasym® device with electrodes on the left earlobe (non-vagal area). Same schedule as active tVNS, combined with Khymeia rehabilitation.
  Arms: Khymeia + Sham tVNS
Device: Traditional Rehabilitation + Active tVNS — Active tVNS with Parasym® (left tragus, 25 Hz, 250 µs, 60 min/day, 5 days/week for 4 weeks) combined with traditional rehabilitation.
  Arms: Traditional Rehabilitation + Active tVNS
Device: Traditional Rehabilitation + Sham tVNS — Sham tVNS with Parasym® device, electrodes on left earlobe, 60 minutes/day, 5 days/week for 4 week. Same duration and schedule, combined with traditional rehabilitation.
  Arms: Traditional Rehabilitation + Sham tVNS

SUMMARY:
This randomized pilot clinical study aims to investigate the effects of trans-auricular vagus nerve stimulation (tVNS) on neuromotor recovery in patients in the subacute phase after stroke. Participants admitted for intensive rehabilitation at ICS Maugeri Centers (Montescano, Pavia, Nervi) will be randomized into four groups receiving either traditional or technological rehabilitation (Khymeia device), combined with active or sham tVNS.

The Parasym® device (CE 0197) delivers non-invasive stimulation of the auricular branch of the vagus nerve at the left ear for 60 minutes daily.

The primary outcome is the improvement in upper limb motor function, assessed by the Fugl-Meyer scale. Secondary outcomes include other clinical, cognitive, and psychological measures, as well as neurophysiological and cardiovascular autonomic parameters.

The study hypothesizes that coupling tVNS with rehabilitation enhances cortical plasticity and accelerates motor recovery. Adverse effects are expected to be minimal, with previous studies reporting only mild transient skin irritation. The results may provide new insights into the neurophysiological mechanisms of recovery and support the integration of non-invasive neuromodulation in post-stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemiplegia following ischemic or hemorrhagic stroke occurred within the previous 6 months, clinically stable
* Age ≥ 18 years
* Single cortical or subcortical lesion documented on neuroimaging, corresponding to the motor deficit
* Cognitively able to understand and follow therapeutic instructions
* Upper limb weakness confirmed by a Motricity Index score below maximum
* Spasticity, if present, compatible with limb function (Modified Ashworth Scale ≤ 2)
* Written informed consent provided

Exclusion Criteria:

* Multiple brain lesions on neuroimaging
* Severe spasticity (Modified Ashworth Scale 3-4)
* Aphasia preventing comprehension of verbal instructions
* Cognitive decline or behavioral disorders interfering with collaboration during training
* Orthopedic conditions or surgical outcomes preventing the execution of the rehabilitation training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-04-03 (Estimated)

PRIMARY OUTCOMES:
Upper limb motor recovery assessed by Fugl-Meyer Assessment (FMA-UE) | Baseline and 4 weeks after treatment

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | Baseline and 4 weeks.
Barthel Index | Baseline and 4 weeks
Mini-Mental State Examination (MMSE) | Baseline and 4 weeks
Frontal Assessment Battery (FAB) | Baseline and 4 weeks
Psychological Scales (PHQ-9) | Baseline and 4 weeks
Psychological Scales (GAD-7) | Baseline and 4 weeks
Somatosensory Evoked Potentials (Median Nerve) | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri - Montescano, Montescano, Pavia, Italy